CLINICAL TRIAL: NCT05525299
Title: The Effects of a Reminiscence-Based Life Review on Copying With Existential Suffering Among Older Cancer Survivors With Cognitive Impairment
Brief Title: Reminiscence-Based Life Review on Copying With Existential Suffering Among Older Cancer Survivors
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Mu-Hsing Ho, Research Assistant Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: uhongkongw4fgupp4
Record Dates: First submitted 2022-08-26; First posted 2022-09-01 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Existential Suffering; Meaning of Life; Cognitive Function; Psychological Distress; Social Support

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): A brief reminiscence-based life review with six themes to recall subjects' memory through the life review reminiscence intervention will be given. A total of six reminiscence chatting sessions (30-60 minutes per session) covering these themes will be conducted weekly.
  Interventions: Behavioral: Reminiscence-Based Life Review
- Control (No Intervention): The subjects allocated in the Control group will not receive any intervention.

INTERVENTIONS:
Behavioral: Reminiscence-Based Life Review — The reminiscence chatting activities covering 6 themes include:
  Week 1: "Instruction of the 'Life Story Narrative Journal' and My 'Childhood' memories" Week 2: "My 'Adolesces' memories and Memorable moments spent with my family" Week 3: "My 'Adulthood' memories and My very first full time job" Week 4: "My thoughts when I received my cancer diagnosis" Week 5: "My favourite activities before and after receiving a cancer diagnosis" Week 6: "When COVID-19 hits, _____ changes and The story goes on! The future pages are more to come!"
  A 'Life Story Narrative Journal' with six themes to recall subjects' memory through the life review reminiscence activities will be given. The Life Story Narrative Journal is a diary booklet that enables the participant to write down and express their thoughts in a narrative.
  Arms: Intervention

SUMMARY:
Target Issue:

Cognitive impairment in older cancer survivors is highly prevalent and the co-existing neuro-psychiatric symptoms, particularly depression, would further complicate the psychosocial consequence of existential suffering. However, no reminiscence-based interventions are specifically developed for older people with cancer have been developed and evaluated.

Target Population:

Cancer survivors aged 65 years old and above with a mild cognitive impairment identified by the HK-MoCA 5-Min Protocol cognitive assessment.

Intervention:

This research project aims to implement a brief reminiscence-based intervention that includes six reminiscence chatting sessions among older cancer survivors. The proposed reminiscence-based intervention has great potential to provide psychological and spiritual care as well as comfort to those who are weak, aged and are in need of assistance.

Study Objectives:

1. To evaluate the effect of a reminiscence-based life review intervention on copying with existential suffering including meaning of life (primary outcome), cognitive function, psychological distress and social support (secondary outcomes) in older cancer survivors
2. To explore older cancer survivors' experience of the intervention regarding the impact of the intervention on their existential suffering

Study Method:

The investigator will recruit 116 voluntary elder patients from the outpatient oncology clinics of the Queen Mary Hospital to participate in the study. They will be individually randomized at a 1:1 ratio to receive usual care or the brief reminiscence-based intervention at home. Outcomes will be assessed at baseline (T0), post-intervention (T1), and 6-week follow-up (T2). A qualitative interview regarding the feedback on the intervention will be undertaken only in the intervention group.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥ 65 years
* Diagnosed with stage I-III non-metastatic cancer
* Completed primary treatment with curative intent (surgery, chemotherapy, and/or radiation therapy) 6 months to 5 years prior to baseline assessments with no recurrence or occurrence of additional cancers
* identified as mild cognitive impairment by the HK-MoCA 5-Min Protocol cognitive assessment (≤ 7th age and education corrected percentile cutoff score)

Exclusion Criteria:

* Inadequate written and verbal Cantonese and/or English comprehension for study activities
* Diagnosed with dementia

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 116 (Estimated)
Dates: Start 2022-10-30 (Actual); Primary Completion 2023-08-30 (Estimated); Study Completion 2024-08-30 (Estimated)

PRIMARY OUTCOMES:
Purpose in life | up to 6 weeks
  The purpose in life will be assessed by the Purpose in Life (PIL) Test developed by Crumbaugh and Maholick (1964), which considers the meaning of life as unique and personal for each individual and as changing throughout the life cycle. The PIL test consists of 20 items that saturate four dimensions: perception of meaning (motives, reasons, and valuation of living life); experience of meaning (perception of one's own life and daily life as full of good things); goals and tasks (goals linked to concrete actions in life and perception of personal responsibility) and dialectic/destiny and freedom (tension between destiny and freedom and coping with death as an uncontrollable, unpredictable, and inevitable event).

SECONDARY OUTCOMES:
Cognitive function | up to 6 weeks
  The objective cognitive function will be assessed by the HK-MoCA 5-Min Protocol cognitive assessment. The HK-MoCA 5-Min Protocol includes four subtests examining five cognitive domains, namely attention, verbal learning and memory, executive functions/language, and orientation. This measure can be alternatively done by a telephone interview and has excellent test-retest reliability, as well as highly correlated with original MoCA. The self-reported cognitive function will be assessed by the FACT-Cog (Functional Assessment of Cancer Therapy - Cognitive Function) scale which consists of 37 items for detecting cancer-related cognitive impairment.
Psychological distress | up to 6 weeks
  The 21-item version of the Depression, Anxiety and Stress Scale (DASS-21) was used to assess mental well-being via core symptoms of depression, anxiety and stress. Each subscale consists of seven self-report items that are each rated on a 4-point self-report scale from 0 (did not apply to me at all) to 3 (applied to me very much, or most of the time). The subscales possess very good psychometric properties in an older population.
Perceived social support | up to 6 weeks
  MSPSS (Multidimensional Scale of Perceived Social Support): 12 items; Likert scale

CONTACTS AND LOCATIONS:
Overall Officials: Mu-Hsing Ho, PhD, Principal Investigator — The University of Hong Kong
Locations (1):
- School of Nursing, The University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided